CLINICAL TRIAL: NCT04689685
Title: The RADAR Study - Wearable-Based Dysglycemia Detection and Warning in Diabetes
Acronym: RADAR
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: ETH Zurich (Other); University of St.Gallen (Other)
Responsible Party: Sponsor
Other Study IDs: RADAR
Record Dates: First submitted 2020-12-24; First posted 2020-12-30 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-09

CONDITIONS: Diabetes Mellitus, Insulin-Dependent; Diabetes
Keywords: Smartwatch; Wearable; Physiological data; Prediction; Dysglycemia; Hyperglycemia; Hypoglycemia
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus; Hyperglycemia; Hypoglycemia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Wearing smartwatch and continous glucose sensor — Patients will be wearing a smartwatch and a continuous glucose meter (CGM) over a maximum duration of 3 months in an outpatient setting.

SUMMARY:
The study RADAR aims at developing a wearable based dysglycemia detection and warning system for patients with diabetes mellitus using artificial intelligence.

DETAILED DESCRIPTION:
Prior research has investigated the general potential of data analytics and artificial intelligence to infer blood glucose levels from a variety of data sources. In this study patients with insulin-dependent diabetes mellitus will be wearing a continuous glucose meter (CGM) and a smartwatch for a maximum duration of 3 months in an outpatient setting. The gathered data will be used to develop a non-invasive and wearable based dysglycemia detection and warning system using artificial intelligence.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent as documented by signature
* Age ≥ 18 years
* Diabetes mellitus treated with multiple daily insulin injections (MDI) or continuous subcutaneous insulin infusion (CSII)

Exclusion Criteria:

* Smartwatch cannot be attached around the wrist of the patient
* Known allergies to components of the Garmin smartwatch or the Dexcom G6 system
* Pregnancy, intention to become pregnant or breast feeding
* Cardiac arrhythmia (e.g. atrial flutter or fibrillation, AV-reentry tachycardia, AV-block > grade 1)
* Pacemaker or ICD (implantable cardioverter defibrillator)
* Treatment with antiarrhythmic drugs or beta-blockers
* Drug or alcohol abuse
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant
* Physical or psychological disease likely to interfere with the normal conduct of the study and interpretation of the study results as judged by the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with insulin-dependent diabetes mellitus treated with multiple daily insulin injections or continuous subcutaneous insulin infusion
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2021-02-19 (Actual); Primary Completion 2022-03-28 (Actual); Study Completion 2022-03-28 (Actual)

PRIMARY OUTCOMES:
Accuracy of the RADAR model: Diagnostic accuracy of wearable based physiological data in detecting dysglycemia (glucose > 13.9mmol/L and glucose < 3.9 mmol/L) quantified as the area under the receiver operator characteristics curve (AUC-ROC) | 4-12 weeks
  Accuracy of the RADAR-model will be assessed using machine learning technology and physiological data recorded by the smartwatch compared to continuous glucose measurements (ground truth)

SECONDARY OUTCOMES:
Accuracy of the RADAR model: Diagnostic accuracy of wearable based physiological data in detecting hypoglycemia (glucose < 3.9 mmol/L) quantified as AUC-ROC | 4-12 weeks
  Accuracy of the RADAR-model will be assessed using machine learning technology and physiological data recorded by the smartwatch compared to continuous glucose measurements (ground truth)
Accuracy of the RADAR model: Diagnostic accuracy of wearable based physiological data in detecting severe hypoglycemia (glucose < 3.0 mmol/L) quantified as AUC-ROC | 4-12 weeks
  Accuracy of the RADAR-model will be assessed using machine learning technology and physiological data recorded by the smartwatch compared to continuous glucose measurements (ground truth)
Accuracy of the RADAR model: Diagnostic accuracy of wearable based physiological data in detecting severe hyperglycemia (glucose > 13.9mmol/L) quantified as AUC-ROC | 4-12 weeks
  Accuracy of the RADAR-model will be assessed using machine learning technology and physiological data recorded by the smartwatch compared to continuous glucose measurements (ground truth)
Accuracy of the RADAR+model: Diagnostic accuracy of wearable based data (physiological, time, fasting glucose, and motion) in detecting dysglycemia (glucose > 13.9mmol/L and glucose < 3.9 mmol/L) quantified as AUC-ROC | 4-12 weeks
  Accuracy of the RADAR+-model will be assessed using machine learning technology and wearable based data (physiological, time, fasting glucose, and motion) compared to continuous glucose measurements (ground truth)
Accuracy of the RADAR+model: Diagnostic accuracy of wearable based data (physiological, time, fasting glucose, and motion) in detecting hypoglycemia (glucose < 3.9 mmol/L) quantified as AUC-ROC | 4-12 weeks
  Accuracy of the RADAR+-model will be assessed using machine learning technology and wearable based data (physiological, time, fasting glucose, and motion) compared to continuous glucose measurements (ground truth)
Accuracy of the RADAR+model: Diagnostic accuracy of wearable based data (physiological, time, fasting glucose, and motion) in detecting severe hypoglycemia (glucose < 3.0 mmol/L) quantified as AUC-ROC | 4-12 weeks
  Accuracy of the RADAR+-model will be assessed using machine learning technology and wearable based data (physiological, time, fasting glucose, and motion) compared to continuous glucose measurements (ground truth)
Accuracy of the RADAR+ model: Diagnostic accuracy of wearable based data (physiological, time, fasting glucose, and motion) in detecting severe hyperglycemia (glucose > 13.9mmol/L) quantified as AUC-ROC | 4-12 weeks
  Accuracy of the RADAR+-model will be assessed using machine learning technology and wearable based data (physiological, time, fasting glucose, and motion) compared to continuous glucose measurements (ground truth)
Accuracy of RADAR-forecast model: Diagnostic accuracy of CGM data in combination with wearable based data (physiological, time, fasting glucose, and motion) in forecasting glucose levels quantified as the mean absolute error. | 4-12 weeks
  Accuracy of the RADAR forecasts will be assessed using machine learning technology, historical continuous glucose measurements data, and historical wearable based data (physiological, time, fasting glucose, and motion) compared to future continuous glucose measurements (ground truth).
Accuracy of the RADAR-forecast model: Diagnostic accuracy of CGM data in combination with wearable based data (physiological, time, fasting glucose, and motion) in forecasting dysglycemia (glucose>13.9mmol/L and glucose<3.9 mmol/L) quantified as AUC-ROC | 4-12 weeks
  Accuracy of the RADAR forecasts will be assessed using machine learning technology, historical continuous glucose measurements data, and historical wearable based data (physiological, time, fasting glucose, and motion) compared to future continuous glucose measurements (ground truth).
Accuracy of the RADAR-forecast model: Diagnostic accuracy of CGM data in combination with wearable based data (physiological, time, fasting glucose, and motion) in forecasting severe hyperglycemia (glucose > 13.9mmol/L) quantified as AUC-ROC | 4-12 weeks
  Accuracy of the RADAR forecasts will be assessed using machine learning technology, historical continuous glucose measurements data, and historical wearable based data (physiological, time, fasting glucose, and motion) compared to future continuous glucose measurements (ground truth).
Accuracy of the RADAR-forecast model: Diagnostic accuracy of CGM data in combination with wearable based data (physiological, time, fasting glucose, and motion) in forecasting mild hypoglycemia (glucose < 3.9mmol/L) quantified as AUC-ROC | 4-12 weeks
  Accuracy of the RADAR forecasts will be assessed using machine learning technology, historical continuous glucose measurements data, and historical wearable based data (physiological, time, fasting glucose, and motion) compared to future continuous glucose measurements (ground truth).
Accuracy of the RADAR-forecast model: Diagnostic accuracy of CGM data in combination with wearable based data (physiological, time, fasting glucose, and motion) in forecasting severe hyperglycemia (glucose < 3.0mmol/L) quantified as AUC-ROC. | 4-12 weeks
  Accuracy of the RADAR forecasts will be assessed using machine learning technology, historical continuous glucose measurements data, and historical wearable based data (physiological, time, fasting glucose, and motion) compared to future continuous glucose measurements (ground truth).
Change of sleep pattern in dysglycemia (< 3.9 mmol/l and > 13.9 mmol/l) compared to eugylcemia. | 4-12 weeks
  Sleep pattern will be recorded by the smartwatch and glucose values are measured with the continuous glucose meter (CGM).
Change of heart rate in dysglycemia (< 3.9 mmol/l and > 13.9 mmol/l) compared to eugylcemia. | 4-12 weeks
  Heart rate will be recorded by the smartwatch and glucose values are measured with the continuous glucose meter (CGM).
Change of heart rate variability (< 3.9 mmol/l and > 13.9 mmol/l) compared to eugylcemia. | 4-12 weeks
  Heart rate variability will be recorded by the smartwatch and glucose values are measured with the continuous glucose meter (CGM).
Change of skin temperature (< 3.9 mmol/l and > 13.9 mmol/l) compared to eugylcemia. | 4-12 weeks
  Skin temperature will be recorded by the smartwatch and glucose values are measured with the continuous glucose meter (CGM).
Change of electrodermal activity (< 3.9 mmol/l and > 13.9 mmol/l) compared to eugylcemia. | 4-12 weeks
  Electrodermal activity will be recorded by the smartwatch and glucose values are measured with the continuous glucose meter (CGM).
Change of stress level (< 3.9 mmol/l and > 13.9 mmol/l) compared to eugylcemia. | 4-12 weeks
  Stress level will be recorded by the smartwatch and glucose values are measured with the continuous glucose meter (CGM).
Influence of sleep duration on daily time in glycemic target range (3.9 - 10 mmol/L) | 4-12 weeks
  Sleep duration will be recorded by the smartwatch and glucose values are measured with the continuous glucose meter (CGM).
Influence on stress-level on daily time in glycemic target range (3.9 - 10 mmol/L) | 4-12 weeks
  Stress level will be recorded by the smartwatch and glucose values are measured with the continuous glucose meter (CGM).
Influence on activity (number of steps and stairs climbed per day) on daily time in glycemic target range (3.9 - 10 mmol/L) | 4-12 weeks
  Number of steps and stairs climbed per day will be recorded by the smartwatch and glucose values are measured with the continuous glucose meter (CGM).
Influence of movement on daily time in glycemic target range (3.9 - 10.0 mmol/l) | 4-12 weeks
  Movement will be recorded by the smartwatch and glucose values are measured with the continuous glucose meter (CGM).
24. Analysis of user requirements for smartwatch based dysglycemia warning systems | 4-12 weeks
  User requirements for the smartwatch based dysglycemia warning system will be assessed in a semi-quantitative interview.

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Stettler, Prof. MD, Principal Investigator — University of Bern
Locations (1):
- Department of Diabetes, Endocrinology, Nutritional Medicine and Metabolism, Bern, Switzerland

REFERENCES:
- [Derived] Lehmann V, Foll S, Maritsch M, van Weenen E, Kraus M, Lagger S, Odermatt K, Albrecht C, Fleisch E, Zueger T, Wortmann F, Stettler C. Noninvasive Hypoglycemia Detection in People With Diabetes Using Smartwatch Data. Diabetes Care. 2023 May 1;46(5):993-997. doi: 10.2337/dc22-2290. PMID 36805169